CLINICAL TRIAL: NCT07318584
Title: Cefotetan Therapy for Escherichia Coli Bacteremia and Genitourinary Infections: a Prospective Phase II Pilot Study
Brief Title: Cefotetan Therapy for Escherichia Coli Infections
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kristina Bajema, Assistant Professor of Medicine, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00028869
Record Dates: First submitted 2025-12-30; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: E Coli Infection; ESBL Producing E.Coli
Keywords: cefotetan; cephamycin; ESBL producing E. coli; E. coli infection
MeSH Terms: conditions — Escherichia coli Infections | interventions — Cefotetan; Carbapenems; Ertapenem; Meropenem; beta Lactam Antibiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cefotetan (Experimental)
  Interventions: Drug: Cefotetan
- Standard of care antibiotics (Active Comparator)
  Interventions: Drug: Carbapenems; Drug: Beta Lactam Antibiotics

INTERVENTIONS:
Drug: Cefotetan — Minimum 1 dose cefotetan within 24 hours of randomization. Creatinine clearance (CrCl) >30 mL/minute: 2 g IV every 12 hours; CrCl 10-30 mL/minute: 2 g IV every 24 hours; CrCl <10 mL/minute: 2 g IV every 48 hours
  Arms: Cefotetan
Drug: Carbapenems — Preferred antibiotic for ESBL E. coli infections: ertapenem. Minimum 1 dose within 24 hours of randomization.
  Other Names: ertapenem; meropenem
  Arms: Standard of care antibiotics
Drug: Beta Lactam Antibiotics — Beta lactam antibiotics for non-ESBL E. coli infections include preferred ceftriaxone or alternative cephalosporins (cefepime, ceftazidime), penicillins (piperacillin-tazobactam, ampicillin-sulbactam), and carbapenems (ertapenem, meropenem). Minimum 1 dose within 24 hours of randomization.
  Arms: Standard of care antibiotics

SUMMARY:
This pilot study will compare clinical outcomes among patients treated with cefotetan versus standard of care antibiotics for bacteremia or genitourinary infections caused by E. coli. It will also measure cefotetan minimum inhibitory concentration (MIC) distributions and cefotetan trough serum concentrations.

DETAILED DESCRIPTION:
In this single-center pilot trial, we will study the efficacy of cefotetan versus standard of care antibiotic therapy for patients hospitalized at Oregon Health & Science University (OHSU) with bacteremia caused by extended-spectrum β-lactamase-producing (ESBL) and non-ESBL E. coli with a genitourinary source. Participants who consent for enrollment will be randomized 1:1 to receive either cefotetan or standard of care antibiotic therapy for their infection and followed for 30 days to determine clinical outcomes. In addition, we will measure cefotetan MIC distributions among patients with ESBL bloodstream or genitourinary infections. Finally, we will measure cefotetan trough serum concentrations in a subset of enrolled patients with ESBL and non-ESBL E. coli bacteremia who are treated with cefotetan.

ELIGIBILITY:
Inclusion Criteria (clinical cohort):

* Identified within 48 hours of inpatient antibiotic administration for acute illness.
* Patient or legally authorized representative are able to provide informed consent for participation in the study.
* Monomicrobial E. coli bacteremia with a genitourinary source.
* Isolate susceptible to both ertapenem and cefotetan (ESBL infections) or ceftriaxone and cefotetan (non-ESBL infections).

Exclusion Criteria (clinical cohort):

* Allergy to cefotetan.
* History of cephalosporin-associated hemolytic anemia.
* Allergy to ertapenem or meropenem (among patients with ESBL E. coli infections).
* Allergy to ceftriaxone (among patients with non-ESBL E. coli infections). Includes allergy to antibiotics with a similar structure expected to confer cross reactivity to ceftriaxone (cefotaxime, cefpodoxime, ceftazidime).
* Admission within 30 previous days.
* Any bacteremia with the same organism in the previous 90 days.
* Pregnant or breastfeeding.
* Moderately to severely immunocompromised, including solid organ or stem cell transplant, hematologic malignancy, active chemotherapy.
* Admission with neutropenic fever.
* Severe illness, including shock and/or intensive care unit admission.
* Inability to complete at least 72 hours of appropriate parenteral therapy, including at least 1 dose cefotetan for patients randomized to the treatment arm or at least 1 dose of appropriate parenteral therapy following randomization for patients assigned to the standard of care arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Clinical success | From randomization through 30 days.
  Absence of death, recurrent E. coli, bacteremia, or need for antibiotic treatment for recurrent E.coli genitourinary infection.

SECONDARY OUTCOMES:
Cefotetan MIC | Baseline
  Cefotetan MIC from E. coli isolated from blood and/or urine culture
Cefotetan trough | Day 1 through 7
  Cefotetan serum trough obtained from a subset of participants randomized to cefotetan arm

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tamma PD, Heil EL, Justo JA, Mathers AJ, Satlin MJ, Bonomo RA. Infectious Diseases Society of America 2024 Guidance on the Treatment of Antimicrobial-Resistant Gram-Negative Infections. Clin Infect Dis. 2024 Aug 7:ciae403. doi: 10.1093/cid/ciae403. Online ahead of print. PMID 39108079
- [Background] Harris PNA, Tambyah PA, Lye DC, Mo Y, Lee TH, Yilmaz M, Alenazi TH, Arabi Y, Falcone M, Bassetti M, Righi E, Rogers BA, Kanj S, Bhally H, Iredell J, Mendelson M, Boyles TH, Looke D, Miyakis S, Walls G, Al Khamis M, Zikri A, Crowe A, Ingram P, Daneman N, Griffin P, Athan E, Lorenc P, Baker P, Roberts L, Beatson SA, Peleg AY, Harris-Brown T, Paterson DL; MERINO Trial Investigators and the Australasian Society for Infectious Disease Clinical Research Network (ASID-CRN). Effect of Piperacillin-Tazobactam vs Meropenem on 30-Day Mortality for Patients With E coli or Klebsiella pneumoniae Bloodstream Infection and Ceftriaxone Resistance: A Randomized Clinical Trial. JAMA. 2018 Sep 11;320(10):984-994. doi: 10.1001/jama.2018.12163. PMID 30208454
- [Background] Stewart AG, Cottrell K, Henderson A, Vemuri K, Bauer MJ, Paterson DL, Harris PNA. In Vitro Activity of Cefotetan against ESBL-Producing Escherichia coli and Klebsiella pneumoniae Bloodstream Isolates from the MERINO Trial. Microbiol Spectr. 2021 Sep 3;9(1):e0022621. doi: 10.1128/Spectrum.00226-21. Epub 2021 Jul 7. PMID 34232101
- See also: Related Info — https://www.accessdata.fda.gov/drugsatfda_docs/label/2020/065430s009lbl.pdf